CLINICAL TRIAL: NCT00337818
Title: A Long-term, Open, Follow-up of the Immunogenicity and Safety of GlaxoSmithKline Biologicals' HPV-16/18 L1/AS04 Vaccine in Healthy Female Subjects Vaccinated Either Pre- or Post-menarche in the Primary Study
Brief Title: Human Papillomavirus (HPV) Vaccine Consistency and Non-inferiority Trial in Young Adult Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 107476 (M18); 107477 (Other: GSK); 107479 (Other: GSK); 107481 (Other: GSK); NCT00337844 (obsolete NCT alias); NCT00337857 (obsolete NCT alias); NCT00338169 (obsolete NCT alias)
Record Dates: First submitted 2006-06-15; First posted 2006-06-16 (Estimated); Results first posted 2010-03-02 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Papillomavirus Type 16/18 Infection; Cervical Intraepithelial Neoplasia
Keywords: Non-inferiority; Immunogenicity; HPV Vaccine Consistency
MeSH Terms: conditions — Uterine Cervical Dysplasia | interventions — human papillomavirus vaccine, L1 type 16, 18

ARMS (3):
- Cervarix New Process (Experimental): Subjects aged 15 to 25 years received 3 doses (at Months 0, 1 and 6) of Cervarix™ (human papillomavirus [HPV]) produced with the new manufacturing process.
  Interventions: Biological: Cervarix™
- Cervarix Old Process Group (Experimental): Subjects aged 15 to 25 years who received 3 doses (at Months 0, 1 and 6) of Cervarix™ (human papillomavirus [HPV]) produced with the old manufacturing process.
  Interventions: Biological: Cervarix™
- Cervarix Young/Lot 1 Group (Experimental): Subjects aged 10 to 14 years, who received 3 doses (at Months 0, 1 and 6) of Cervarix™ (human papillomavirus [HPV]) produced with the new manufacturing process (Lot 1).
  Interventions: Biological: Cervarix™

INTERVENTIONS:
Biological: Cervarix™ — Three doses of vaccine according to a 0, 1, 6 month schedule (during the primary study)

SUMMARY:
The study will be extended for subjects who received all three doses of vaccine in Finland, Denmark and Estonia to determine long-term safety and immunogenicity of the HPV-16/18 vaccine. Human Papilloma virus (HPV) are viruses that cause a common infection of the skin and genitals in men and women. Several types of HPV infection are transmitted by sexual activity and, in women, can infect the cervix (part of the uterus or womb). This infection often goes away by itself, but if it does not go away (this is called persistent infection), it can lead in women over a long period of time to cancer of the cervix. If a woman is not infected by HPV, it is very unlikely that she will get cervical cancer. This study will evaluate the consistency of consecutive vaccine lots and the non-inferiority of modified manufacturing processes of GlaxoSmithKline Biologicals HPV-16/18 vaccine and the vaccine safety, over 12 months, in young adolescents and women of 10-25 years of age at study start.

DETAILED DESCRIPTION:
Approximately 750 study subjects received different lots of the HPV vaccine administered intramuscularly according to a 0-1-6 month schedule.

The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

ELIGIBILITY:
Inclusion Criteria:

* A female who enrolled in the HPV-012 (NCT00337818) study in Denmark, Estonia and Finland, received three doses of vaccine and completed Visit 4 (Month 7).
* Written informed consent obtained from the subject prior to enrolment (for subjects below the legal age of consent, written informed consent must be obtained from a parent or legally acceptable representative (LAR) and, in addition, the subject must sign and personally date a written informed assent).

Exclusion criteria

* Use of any investigational or non-registered product (drug or vaccine) or planned use during the study period.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).
* Chronic administration of immunosuppressants or other immune-modifying drugs occurring less than three months prior to blood sampling.
* Administration of immunoglobulins and/or any blood products within the three months preceding blood sampling.

Ages: 10 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 770 (Actual)
Dates: Start 2006-06; Primary Completion 2006-06 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Tallinn, Estonia

REFERENCES:
- See also: Primary Study — http://www.clinicaltrials.gov/ct/show/NCT00169494

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Only 8 subjects came to Month 18 whereas most of the subjects came to Month 24. Therefore, no separate analysis at Month 18 was prepared; data for Month 18 outcome variables were incorporated into Month 24 analyses.
Groups:
- Cervarix New Process: Subjects aged 15 to 25 years received 3 doses (at Months 0, 1 and 6) of Cervarix™ (human papillomavirus [HPV] vaccine) produced with the new manufacturing process.
- Cervarix Old Process Group: Subjects aged 15 to 25 years who received 3 doses (at Months 0, 1 and 6) of Cervarix™ (human papillomavirus [HPV] vaccine) produced with the old manufacturing process.
- Cervarix Young: Subjects aged 10 to 14 years, who received 3 doses (at Months 0, 1 and 6) of Cervarix™ (human papillomavirus [HPV] vaccine) produced with the new manufacturing process.
Period: Overall Study
Arm/Group | Cervarix New Process | Cervarix Old Process Group | Cervarix Young
Started | 458 | 154 | 158
Completed | 169 | 63 | 51
Not Completed | 289 | 91 | 107
Not completed — Lost to Follow-up | 289 | 91 | 107

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cervarix New Process | Cervarix Old Process Group | Cervarix Young | Total
Number analyzed (Participants) | 458 | 154 | 158 | 770
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.2 (2.96) | 20.3 (2.99) | 12.4 (1.37) | 18.6 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 458 | 154 | 158 | 770
  Male | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Titers of Anti-human Papilloma Virus 16 (Anti-HPV-16) and Anti-human Papilloma Virus 18 (Anti-HPV-18) Antibodies
Description: Titers are given as Geometric Mean Titers (GMTs) expressed as Enzyme-linked Immunosorbent Assay Units Per Milliliter (EL.U/mL).
  *Data for Month 18 outcome variables were incorporated into the Month 24 analyses.
Time Frame: At months 18*, 24, 36 and 48
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for analysis of immunogenicity, on subjects with available data for the defined timepoint.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Cervarix New Process | Cervarix Old Process Group | Cervarix Young
Number analyzed (Participants) | 160 | 51 | 55
EL.U/mL
  Anti-HPV-16 (Month 24) (n=160, 51, 55) | 1440.4 [1249.3 to 1660.7] | 1903.7 [1396.0 to 2596.0] | 3861.7 [2947.0 to 5060.4]
  Anti-HPV-16 (Month 36) (n=150, 46, 52) | 1397.5 [1207.1 to 1618.1] | 1679.3 [1211.5 to 2327.6] | 3353.0 [2553.4 to 4403.1]
  Anti-HPV-16 (Month 48) (n=141, 49, 49) | 1140.9 [974.9 to 1335.3] | 1427.3 [1027.6 to 1982.4] | 2862.2 [2129.3 to 3847.3]
  Anti-HPV-18 (Month 24) (n=160, 50, 54) | 649.8 [554.3 to 761.8] | 778.8 [577.1 to 1050.8] | 1341.8 [1053.2 to 1709.6]
  Anti-HPV-18 (Month 36) (n=151, 45, 51) | 574.7 [490.2 to 673.7] | 649.6 [464.5 to 908.4] | 1111.0 [848.5 to 1454.9]
  Anti-HPV-18 (Month 48) (n=141, 48, 48) | 462.4 [391.5 to 546.1] | 519.9 [374.1 to 722.4] | 935.6 [717.9 to 1219.5]

2. Secondary Outcome: Titers of Anti-human Papilloma Virus 16 (Anti-HPV-16) and Anti-human Papilloma Virus 18 (Anti-HPV-18) Antibodies in Cervical Samples
Description: Titers are given as Geometric Mean Titers (GMTs) expressed as EL.U/mL.
Time Frame: At months 24, 36, and 48
Population: Analysis was performed on the ATP cohort for analysis of immunogenicity, in post-menarcheal subjects who volunteered for cervicovaginal sampling collection and with cervicovaginal secretion samples having less than 80 erythrocytes per milliliter and with results available for the defined timepoint.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Cervarix New Process | Cervarix Old Process Group | Cervarix Young
Number analyzed (Participants) | 78 | 27 | 4
EL.U/mL
  HPV-16 (Month 24) (n= 55, 13, 1) | 85.4 [57.9 to 125.8] | 107.5 [47.5 to 242.8] | 198.8 [198.8 to 198.8]
  HPV-16 (Month 36) (n= 78, 27, 3) | 68.2 [54.6 to 85.2] | 62.1 [40.8 to 94.7] | 63.4 [4.8 to 845.9]
  HPV-16 (Month 48) (n=69, 19, 4) | 56.2 [43.4 to 72.8] | 94.5 [50.8 to 175.8] | 129.2 [12.8 to 1305.0]
  HPV-18 (Month 24) (n= 55, 13, 1) | 45.9 [31.1 to 67.6] | 31.9 [15.8 to 64.4] | 107.9 [107.9 to 107.9]
  HPV-18 (Month 36) (n= 78, 27, 3) | 38.9 [31.2 to 48.6] | 29.6 [19.8 to 44.2] | 19.9 [1.1 to 362.2]
  HPV-18 (Month 48) (n= 66, 19, 4) | 33.9 [24.7 to 46.5] | 48.8 [26.4 to 90.0] | 97.5 [38.7 to 245.4]

3. Secondary Outcome: Titers of Anti-HPV-16 and Anti-HPV-18 Immunoglobulin G (IgG) Antibodies in Blood Samples
Description: Titers are given as Geometric Mean Titers (GMTs) expressed as EL.U/mL.
Time Frame: At Months 24, 36 and 48
Population: Analysis was performed on the Total Vaccinated Cohort, on subjects with cervicovaginal secretion sample results available and with cervicovaginal secretion samples having less than 200 erythrocytes per milliliter and with results available for the defined timepoint.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Cervarix New Process | Cervarix Old Process Group | Cervarix Young
Number analyzed (Participants) | 78 | 27 | 4
EL.U/mL
  Anti-HPV-16 [Month 24] (n=74;24;3) | 1403.1 [1126.9 to 1747.0] | 1490.5 [1016.1 to 2186.5] | 5399.5 [367.9 to 79243.9]
  Anti-HPV-16 [Month 36] (n=78;27;3) | 1291.8 [1030.9 to 1618.7] | 1435.0 [993.0 to 2073.8] | 3733.3 [383.1 to 36384.7]
  Anti-HPV-16 [Month 48] (n=69;19;4) | 1047.3 [854.2 to 1284.0] | 1950.5 [1095.1 to 3474.1] | 3332.7 [1087.6 to 10212.5]
  Anti-HPV-18 [Month 24] (n=74;24;3) | 584.5 [461.1 to 741.0] | 648.6 [467.7 to 899.6] | 1814.6 [240.3 to 13702.9]
  Anti-HPV-18 [Month 36] (n=78;27;3) | 555.4 [439.3 to 702.1] | 542.1 [392.8 to 748.0] | 1163.6 [88.8 to 15244.0]
  Anti-HPV-18 [Month 48] (n=66;19;4) | 478.4 [376.8 to 607.3] | 805.4 [491.2 to 1320.5] | 1048.9 [250.5 to 4392.8]

4. Secondary Outcome: Number of Subjects Reporting Pregnancies, New Onset Chronic Diseases (NOCDs) and Other Medically Significant Conditions (MSCs)
Description: NOCDs assessed include e.g. autoimmune disorders, asthma, type I diabetes. MSCs assessed include adverse events prompting emergency room or physician visits that are not related to common diseases or serious adverse events (SAEs) that are not related to common diseases.
Time Frame: Throughout the study period (up to Month 48)
Population: Analysis was performed on the Total vaccinated cohort for Month 24, Month 36 and Month 48, respectively.
Measure: Number; unit: Subjects
Arm/Group | Cervarix New Process | Cervarix Old Process Group | Cervarix Young
Number analyzed (Participants) | 186 | 65 | 57
Subjects
  NOCDs from Month 12 to Month 24 (n= 186, 64, 57) | 1 | 0 | 1
  NOCDs from Month 24 to Month 36 (n= 184, 65, 53) | 3 | 0 | 1
  NOCDs from Month 36 to Month 48 (n= 169, 63, 51) | 0 | 1 | 1
  MSCs from Month 12 to Month 24 (n= 186, 64, 57) | 12 | 4 | 2
  MSCs from Month 24 to Month 36 (n= 184, 65, 53) | 35 | 10 | 6
  MSCs from Month 36 to Month 48 (n= 169, 63, 51) | 19 | 5 | 1
  Pregnancies from Month 12 to Month 24(n=186,64,57) | 4 | 2 | 0
  Pregnancies from Month 24 to Month 36(n=184,65,53) | 20 | 7 | 0
  Pregnancies from Month 36 to Month 48(n=169,63,51) | 15 | 6 | 1

5. Secondary Outcome: Number of Subjects Reporting SAEs
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: Throughout the study period (up to Month 48)
Population: Analysis was performed on the Total vaccinated cohort of each time point.
Measure: Number; unit: Subjects
Arm/Group | Cervarix New Process | Cervarix Old Process Group | Cervarix Young
Number analyzed (Participants) | 186 | 65 | 57
Subjects
  From Month 12 to 24 (n=186,64,57) | 2 | 1 | 0
  From Month 24 to 36 (n=184,65,53) | 7 | 0 | 3
  From Month 36 to 48 (n=169,63,51) | 5 | 2 | 0

ADVERSE EVENTS:
Time Frame: During the entire long-term follow-up of the study: data collected at Month 18, 24, 36 and 48.
Description: Other (non-serious) adverse event data were not collected in the framework of this long-term follow-up study.
  The number of subjects at risk for each individal adverse event corresponds to the total number of subjects included in the total vaccinated cohort of the particular timepoint at which the adverse event was reported.
Arm/Group | Cervarix New Process | Cervarix Old Process Group | Cervarix Young
Serious Adverse Events (participants affected / at risk) | 11/186 | 3/65 | 3/57
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Cervarix New Process (N=186) | Cervarix Old Process Group (N=65) | Cervarix Young (N=57)
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Anogenital warts (Infections and infestations) | 1 | 0 | 0
Enteritis infectious (Infections and infestations) | 1 | 0 | 0
Genital herpes (Infections and infestations) | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blighted ovum (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Endometriosis (Reproductive system and breast disorders) | 2 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0/169 | 2/63 | 0/51
Chorioamnionitis (Pregnancy, puerperium and perinatal conditions) | 1/169 | 0/63 | 0/51
Diarrhoea (Gastrointestinal disorders) | 1/169 | 0/63 | 0/51
Enterocolitis infectious (Infections and infestations) | 1/169 | 0/63 | 0/51
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 1/169 | 0/63 | 0/51
Pyelonephritis (Infections and infestations) | 0 | 1/64 | 0
Premature separation of placenta (Pregnancy, puerperium and perinatal conditions) | 1 | 0/64 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0/64 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.